CLINICAL TRIAL: NCT06103513
Title: A Randomized Clinical Trial of Two Different Initial Growth Hormone Doses in Children With Growth Hormone Deficiency in the First Year of Treatment
Brief Title: Randomized Clinical Trial of Two Different Initial Growth Hormone Doses in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-0027
Record Dates: First submitted 2023-10-17; First posted 2023-10-26 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-10

CONDITIONS: Growth Disorders; Growth Failure; Growth Hormone Treatment; Growth
Keywords: Growth Hormone
MeSH Terms: conditions — Growth Disorders; Failure to Thrive | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Growth hormone 0.2 mg/kg/week (Active Comparator): Twenty-five subjects will initiate rhGH therapy at 0.2 mg/kg/week for the first 12 months of treatment
  Interventions: Drug: Somatropin
- Arm 2: Growth hormone 0.3 mg/kg/week (Active Comparator): Twenty-five subjects will initiate rhGH therapy at 0.3 mg/kg/week for the first 12 months of treatment
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — The treatment of children with subcutaneous recombinant human growth hormone (rhGH) is the current gold standard of care for children with diagnosed GHD. This study will serve only to investigate the optimal dose of treatment in the first year of treatment with rhGH.
  Other Names: Norditropin, Nutropin AQ, Genotropin, Zomacton, Humatrope, Omnitrope.

SUMMARY:
A prospective, randomized, open-label single-blinded study of 50 subjects with growth hormone deficiency, ages 5 to 15 years in which 25 subjects will initiate rhGH therapy at 0.3mg/kg/week and the remaining 25 subjects will initiate their rhGH treatment at 0.2 mg/kg/week for the first 12 months of treatment. Safety parameters, height velocity, and adult height prediction by bone age determination will be assessed at 4-month intervals for 1 year following the initiation of rhGH therapy.

DETAILED DESCRIPTION:
Investigators propose a prospective randomized, open-label single-blinded study of 50 subjects with growth hormone deficiency, ages 5 to 15 years. 25 subjects will be randomized to initiate a dose of 0.3 mg/kg/week (0.28-0.32 mg/kg/week) and the remaining 25 subjects will initiate their rhGH treatment at 0.2 mg/kg/week (0.18-0.22 mg/kg/week) for the first 12 months of treatment. Safety parameters, height velocity, and adult height prediction by bone age determination will be assessed at 4-month intervals for 1 year following the initiation of rhGH therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 5-15 years
4. In good general health as evidenced by medical history or diagnosed with growth hormone deficiency
5. Ability to take subcutaneous GH injections nightly

Exclusion Criteria:

Subjects will be excluded if they have GH resistance, or syndromic short stature such as Prader Willi syndrome and Turner syndrome. Patients will also be excluded if they have active malignancies, or systemic illnesses such as heart failure, kidney failure, or liver failure.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Annualized Growth Velocity (GV) in the first year after treatment | I year
  Height (cm) at 0- month visit; height (cm) at 12-month visit

SECONDARY OUTCOMES:
IGF1- 0,4,8,12 months | 12 Months
  IGF-1 will be collected at timepoints - 0,4,8,12 months
IGFBP3 - 0,4,8,12 months | 12 Months
  IGFBP3 will be collected at timepoints - 0,4,8,12 months
HbA1c - 4,8,12 months | 12 Months
  HbA1c will be collected at timepoints 4,8,12 months
Total T4 or Free T4 - 0,12 months | 12 Months
  Total T4 or Free T4 will be collected at timepoints 0,12 months
TSH - 0, 12 months | 12 Months
  TSH will be collected at timepoints 0, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin U. Nwosu, MD, Principal Investigator — NORTHWELL HEALTH, INC.
Locations (1):
- Northwell Health, New York, New York, United States

REFERENCES:
- [Background] Backelijaw P, Dattani M, Cohen P Rosenfeld R, (2014).Chapter 10: Disorders of Growth Hormone/ Insulin Like Growth Factor Secretion and Action. Shreiner, J (Ed.). Pediatric Endocrinology: Marc Sperling. (chapter 10, page 364, 366). Philadelphia, Saunders
- [Background] Grumbach MM, Bin-Abbas BS, Kaplan SL. The growth hormone cascade: progress and long-term results of growth hormone treatment in growth hormone deficiency. Horm Res. 1998;49(# Suppl 2):41-57. No abstract available. PMID 9716827
- [Background] Blethen SL, MacGillivray MH. A risk-benefit assessment of growth hormone use in children. Drug Saf. 1997 Nov;17(5):303-16. doi: 10.2165/00002018-199717050-00003. PMID 9391774
- [Background] Christ ER, Cummings MH, Jackson N, Stolinski M, Lumb PJ, Wierzbicki AS, Sonksen PH, Russell-Jones DL, Umpleby AM. Effects of growth hormone (GH) replacement therapy on low-density lipoprotein apolipoprotein B100 kinetics in adult patients with GH deficiency: a stable isotope study. J Clin Endocrinol Metab. 2004 Apr;89(4):1801-7. doi: 10.1210/jc.2003-031474. PMID 15070948
- [Background] Locatelli V, Bianchi VE. Effect of GH/IGF-1 on Bone Metabolism and Osteoporsosis. Int J Endocrinol. 2014;2014:235060. doi: 10.1155/2014/235060. Epub 2014 Jul 23. PMID 25147565
- [Background] Boguszewski CL, Meister LH, Zaninelli DC, Radominski RB. One year of GH replacement therapy with a fixed low-dose regimen improves body composition, bone mineral density and lipid profile of GH-deficient adults. Eur J Endocrinol. 2005 Jan;152(1):67-75. doi: 10.1530/eje.1.01817. PMID 15762189
- [Background] Hardin DS. Treatment of short stature and growth hormone deficiency in children with somatotropin (rDNA origin). Biologics. 2008 Dec;2(4):655-61. doi: 10.2147/btt.s2252. PMID 19707446
- [Background] Straetemans S, Thomas M, Craen M, Rooman R, De Schepper J; BESPEED. Poor growth response during the first year of growth hormone treatment in short prepubertal children with growth hormone deficiency and born small for gestational age: a comparison of different criteria. Int J Pediatr Endocrinol. 2018;2018:9. doi: 10.1186/s13633-018-0064-3. Epub 2018 Oct 22. PMID 30377433
- [Background] Reiter EO, Price DA, Wilton P, Albertsson-Wikland K, Ranke MB. Effect of growth hormone (GH) treatment on the near-final height of 1258 patients with idiopathic GH deficiency: analysis of a large international database. J Clin Endocrinol Metab. 2006 Jun;91(6):2047-54. doi: 10.1210/jc.2005-2284. Epub 2006 Mar 14. PMID 16537676
- [Background] de Ridder MA, Stijnen T, Hokken-Koelega AC. Prediction of adult height in growth-hormone-treated children with growth hormone deficiency. J Clin Endocrinol Metab. 2007 Mar;92(3):925-31. doi: 10.1210/jc.2006-1259. Epub 2006 Dec 19. PMID 17179199
- [Background] Wit JM, Ranke MB, Albertsson-Wikland K, Carrascosa A, Rosenfeld RG, Van Buuren S, Kristrom B, Schoenau E, Audi L, Hokken-Koelega AC, Bang P, Jung H, Blum WF, Silverman LA, Cohen P, Cianfarani S, Deal C, Clayton PE, de Graaff L, Dahlgren J, Kleintjens J, Roelants M. Personalized approach to growth hormone treatment: clinical use of growth prediction models. Horm Res Paediatr. 2013;79(5):257-70. doi: 10.1159/000351025. Epub 2013 May 28. PMID 23735882
- [Background] Kristrom B, Dahlgren J, Niklasson A, Nierop AF, Albertsson-Wikland K. The first-year growth response to growth hormone treatment predicts the long-term prepubertal growth response in children. BMC Med Inform Decis Mak. 2009 Jan 12;9:1. doi: 10.1186/1472-6947-9-1. PMID 19138407
- [Background] MacGillivray MH, Baptista J, Johanson A. Outcome of a four-year randomized study of daily versus three times weekly somatropin treatment in prepubertal naive growth hormone-deficient children. Genentech Study Group. J Clin Endocrinol Metab. 1996 May;81(5):1806-9. doi: 10.1210/jcem.81.5.8626839.
- [Background] Ranke MB, Schweizer R, Wollmann HA, Schwarze P. Dosing of growth hormone in growth hormone deficiency. Horm Res. 1999;51 Suppl 3:70-4. doi: 10.1159/000053165. PMID 10592447
- [Background] Ranke MB, Lindberg A, Chatelain P, Wilton P, Cutfield W, Albertsson-Wikland K, Price DA. Derivation and validation of a mathematical model for predicting the response to exogenous recombinant human growth hormone (GH) in prepubertal children with idiopathic GH deficiency. KIGS International Board. Kabi Pharmacia International Growth Study. J Clin Endocrinol Metab. 1999 Apr;84(4):1174-83. doi: 10.1210/jcem.84.4.5634. PMID 10199749
- [Background] Sudfeld H, Kiese K, Heinecke A, Bramswig JH. Prediction of growth response in prepubertal children treated with growth hormone for idiopathic growth hormone deficiency. Acta Paediatr. 2000 Jan;89(1):34-7. doi: 10.1080/080352500750029022. PMID 10677054
- [Background] Kristrom B, Aronson AS, Dahlgren J, Gustafsson J, Halldin M, Ivarsson SA, Nilsson NO, Svensson J, Tuvemo T, Albertsson-Wikland K. Growth hormone (GH) dosing during catch-up growth guided by individual responsiveness decreases growth response variability in prepubertal children with GH deficiency or idiopathic short stature. J Clin Endocrinol Metab. 2009 Feb;94(2):483-90. doi: 10.1210/jc.2008-1503. Epub 2008 Nov 11. PMID 19001519
- [Background] Radetti G, Buzi F, Paganini C, Pilotta A, Felappi B. Treatment of GH-deficient children with two different GH doses: effect on final height and cost-benefit implications. Eur J Endocrinol. 2003 May;148(5):515-8. doi: 10.1530/eje.0.1480515. PMID 12720533
- [Background] Cho WK, Ahn MB, Kim EY, Cho KS, Jung MH, Suh BK. Predicting First-Year Growth in Response to Growth Hormone Treatment in Prepubertal Korean Children with Idiopathic Growth Hormone Deficiency: Analysis of Data from the LG Growth Study Database. J Korean Med Sci. 2020 May 18;35(19):e151. doi: 10.3346/jkms.2020.35.e151. PMID 32419399